CLINICAL TRIAL: NCT04513613
Title: A Post-Market Registry for the Evaluation of the CorPath® GRX System Effectiveness in Peripheral Vascular Interventions
Brief Title: ACHIEVE GRX Registry
Status: Withdrawn | Type: Observational
Why Stopped: Sites have adjusted their participation priorities due to the pandemic. Not enough site interest at this current time to initiate the study.
Sponsor: Corindus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 104-09200
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases; Renal Artery Disease; Carotid Artery Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with a clinical indication for PVI: Subjects with a clinical indication for Peripheral Vascular Intervention (PVI).
  Interventions: Device: Procedure/Surgery: Robotic-PVI

INTERVENTIONS:
Device: Procedure/Surgery: Robotic-PVI — Robotic-assisted (CorPath GRX System) percutaneous vascular interventions.

SUMMARY:
This study will evaluate real-world performance of the CorPath GRX System in peripheral vascular interventions.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label, multi-center registry of the CorPath GRX System to evaluate its real-world performance during peripheral vascular interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subject has a clinical indication for Peripheral Vascular Intervention (PVI).
3. Subject is deemed appropriate for robotic-assisted PVI.
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
5. Individual monitoring of radiation dose, using the pocket dosimeter, was initiated at start of procedure.

Exclusion Criteria:

1. Failure/inability/unwillingness to provide informed consent.
2. The investigator determines the subject or the peripheral anatomy is not suitable for ro-botic-assisted PVI.
3. Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a clinical indication for Peripheral Vascular Intervention (PVI).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Procedure
  Successful completion of the robotic-assisted endovascular procedure absent any unplanned conversion to manual for guidewire or balloon/stent catheter inability to navigate vessel anatomy.
Clinical Success | Within 24 hours of the procedure or hospital discharge, whichever occurs first.
  <30% residual stenosis in all CorPath System treated lesions at the completion of the interventional procedure in the absence of device-related serious adverse event (SAE).
Safety | Within 24 hours of the procedure or hospital discharge, whichever occurs first.
  A composite of intra- and peri-procedural events, including target vessel rupture, clinically significant perforation or dissection, and distal embolization.

SECONDARY OUTCOMES:
PVI Procedure Time | Procedure
  Defined as the time measured from the insertion of the guiding sheath until the removal of the guiding sheath.
Manual Time | Procedure
  Defined as the total amount of time the procedure is completed using a manual technique.
Robotic Time | Procedure
  Defined as the total amount of time the procedure is completed robotically from the robotic cock-pit.
Fluoroscopy Time | Procedure
  Total fluoroscopy utilized during the procedure as recorded by an Imaging System.
Operator Radiation Exposure | Procedure
  Cumulative dose the operator receives as recorded from an electronic pocket dosimeter during the procedure.
Staff Radiation Exposure | Procedure
  Cumulative dose the staff receives as recorded from an electronic pocket dosimeter during the procedure.
Patient Radiation Exposure | Procedure
  DAP (dose-area-product) and AK (air kerma) as recorded during the procedure.
Contrast Fluid Volume | Procedure
  Total volume of contrast (mL) used during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jon George, MD, Principal Investigator — Einstein Medical Center; John Phillips, MD, Principal Investigator — Riverside Methodist Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Dijk LJ, van Noord D, de Vries AC, Kolkman JJ, Geelkerken RH, Verhagen HJ, Moelker A, Bruno MJ. Clinical management of chronic mesenteric ischemia. United European Gastroenterol J. 2019 Mar;7(2):179-188. doi: 10.1177/2050640618817698. Epub 2018 Dec 4. PMID 31080602
- [Background] Uccioli L, Meloni M, Izzo V, Giurato L, Merolla S, Gandini R. Critical limb ischemia: current challenges and future prospects. Vasc Health Risk Manag. 2018 Apr 26;14:63-74. doi: 10.2147/VHRM.S125065. eCollection 2018. PMID 29731636
- [Background] Dalal PK, Prasad A. Contemporary Outcomes of Endovascular Intervention for Critical Limb Ischemia. Interv Cardiol Clin. 2017 Apr;6(2):251-259. doi: 10.1016/j.iccl.2016.12.008. Epub 2017 Jan 27. PMID 28257772
- [Background] Canfield J, Totary-Jain H. 40 Years of Percutaneous Coronary Intervention: History and Future Directions. J Pers Med. 2018 Oct 1;8(4):33. doi: 10.3390/jpm8040033. PMID 30275411
- [Background] Benjamin R, Lui F. Vertebrobasilar Insufficiency. 2025 Dec 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482259/ PMID 29489229
- [Background] Schoepe R, McQuillan S, Valsan D, Teehan G. Atherosclerotic Renal Artery Stenosis. Adv Exp Med Biol. 2017;956:209-213. doi: 10.1007/5584_2016_89. PMID 27873231
- [Background] Writing Committee Members; Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FGR, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RAG, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME; ACC/AHA Task Force Members; Halperin JL, Levine GN, Al-Khatib SM, Birtcher KK, Bozkurt B, Brindis RG, Cigarroa JE, Curtis LH, Fleisher LA, Gentile F, Gidding S, Hlatky MA, Ikonomidis J, Joglar J, Pressler SJ, Wijeysundera DN. 2016 AHA/ACC Guideline on the Management of Patients with Lower Extremity Peripheral Artery Disease: Executive Summary. Vasc Med. 2017 Jun;22(3):NP1-NP43. doi: 10.1177/1358863X17701592. No abstract available. PMID 28494710
- [Background] White RD, Weir-McCall JR, Sullivan CM, Mustafa SA, Yeap PM, Budak MJ, Sudarshan TA, Zealley IA. The celiac axis revisited: anatomic variants, pathologic features, and implications for modern endovascular management. Radiographics. 2015 May-Jun;35(3):879-98. doi: 10.1148/rg.2015140243. Epub 2015 Apr 17. PMID 25884099
- [Background] Beckman JA, Creager MA. Chapter 18 Peripheral Artery Disease Clinical Evaluation. In: Creager MA, Beckman JA, Loscalzo J, eds. Vascular Medicine: A Companion to Braunwald's Heart Disease. Philadelphia, PA: Elsevier Saunders; 2013
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883
- [Background] Allison MA, Ho E, Denenberg JO, Langer RD, Newman AB, Fabsitz RR, Criqui MH. Ethnic-specific prevalence of peripheral arterial disease in the United States. Am J Prev Med. 2007 Apr;32(4):328-33. doi: 10.1016/j.amepre.2006.12.010. PMID 17383564
- [Background] Klein LW, Miller DL, Balter S, Laskey W, Haines D, Norbash A, Mauro MA, Goldstein JA; Joint Inter-Society Task Force on Occupational Hazards in the Interventional Laboratory. Occupational health hazards in the interventional laboratory: time for a safer environment. Catheter Cardiovasc Interv. 2009 Feb 15;73(3):432-8. doi: 10.1002/ccd.21801. PMID 19214981
- [Background] Kim KP, Miller DL, Balter S, Kleinerman RA, Linet MS, Kwon D, Simon SL. Occupational radiation doses to operators performing cardiac catheterization procedures. Health Phys. 2008 Mar;94(3):211-27. doi: 10.1097/01.HP.0000290614.76386.35. PMID 18301095
- [Background] Vano E, Gonzalez L, Beneytez F, Moreno F. Lens injuries induced by occupational exposure in non-optimized interventional radiology laboratories. Br J Radiol. 1998 Jul;71(847):728-33. doi: 10.1259/bjr.71.847.9771383.
- [Background] Goldsweig AM, Abbott JD, Aronow HD. Physician and Patient Radiation Exposure During Endovascular Procedures. Curr Treat Options Cardiovasc Med. 2017 Feb;19(2):10. doi: 10.1007/s11936-017-0507-9. PMID 28275940
- [Background] El-Sayed T, Patel AS, Cho JS, Kelly JA, Ludwinski FE, Saha P, Lyons OT, Smith A, Modarai B; Guy's and St Thomas' Cardiovascular Research Collaborative. Radiation-Induced DNA Damage in Operators Performing Endovascular Aortic Repair. Circulation. 2017 Dec 19;136(25):2406-2416. doi: 10.1161/CIRCULATIONAHA.117.029550. Epub 2017 Oct 20. PMID 29054934
- [Background] Goldsweig AM, Kennedy KF, Kolte D, Abbott JD, Gordon PC, Sharaf BL, Sellke FW, Ehsan A, Sodha NR, Rutar F, Aronow HD. Predictors of patient radiation exposure during transcatheter aortic valve replacement. Catheter Cardiovasc Interv. 2018 Oct 1;92(4):768-774. doi: 10.1002/ccd.27452. Epub 2017 Dec 27. PMID 29280551
- [Background] Mahmud E, Schmid F, Kalmar P, Deutschmann H, Hafner F, Rief P, Brodmann M. Feasibility and Safety of Robotic Peripheral Vascular Interventions: Results of the RAPID Trial. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2058-2064. doi: 10.1016/j.jcin.2016.07.002. Epub 2016 Sep 14. PMID 27639904
- [Background] Vano E, Gonzalez L, Fernandez JM, Haskal ZJ. Eye lens exposure to radiation in interventional suites: caution is warranted. Radiology. 2008 Sep;248(3):945-53. doi: 10.1148/radiol.2482071800. Epub 2008 Jul 15. PMID 18632529
- [Background] Weisz G, Metzger DC, Caputo RP, Delgado JA, Marshall JJ, Vetrovec GW, Reisman M, Waksman R, Granada JF, Novack V, Moses JW, Carrozza JP. Safety and feasibility of robotic percutaneous coronary intervention: PRECISE (Percutaneous Robotically-Enhanced Coronary Intervention) Study. J Am Coll Cardiol. 2013 Apr 16;61(15):1596-600. doi: 10.1016/j.jacc.2012.12.045. PMID 23500318
- [Background] Smitson CC, Ang L, Pourdjabbar A, Reeves R, Patel M, Mahmud E. Safety and Feasibility of a Novel, Second-Generation Robotic-Assisted System for Percutaneous Coronary Intervention: First-in-Human Report. J Invasive Cardiol. 2018 Apr;30(4):152-156. Epub 2018 Jan 15. PMID 29335386
- [Background] Smilowitz NR, Moses JW, Sosa FA, Lerman B, Qureshi Y, Dalton KE, Privitera LT, Canone-Weber D, Singh V, Leon MB, Weisz G. Robotic-Enhanced PCI Compared to the Traditional Manual Approach. J Invasive Cardiol. 2014 Jul;26(7):318-21. PMID 24993988
- [Background] Mahmud E, Dominguez A, Bahadorani J. First-in-human robotic percutaneous coronary intervention for unprotected left main stenosis. Catheter Cardiovasc Interv. 2016 Oct;88(4):565-570. doi: 10.1002/ccd.26550. Epub 2016 May 18. PMID 27189238

DOCUMENTS (1):
  • Study Protocol (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT04513613/Prot_000.pdf